CLINICAL TRIAL: NCT02347020
Title: Impact of Sleep and Meal Timing on Food Intake Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Assitant Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAO1801; 1R56HL119945 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Diabetes Mellitus, Type II; Cardiovascular Disease
Keywords: Obesity; Metabolic Disorders
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal Sleep/ Normal Meal (Experimental): sleep 0000-0800 h, meals at 1, 5, 11, and 12.5 (snack) h after awakening
  Interventions: Behavioral: Normal Sleep/ Normal Meal
- Normal Sleep/ Late Meal (Experimental): Ns/Lm: sleep 0000-0800 h, meals at 4.5, 8.5, 14.5, and 16 (snack) h after awakening
  Interventions: Behavioral: Normal Sleep/ Late Meal
- Late Sleep/ Normal Meal (Experimental): sleep 0330-1130 h, meals at 1, 5, 11, and 12.5 (snack) h after awakening
  Interventions: Behavioral: Late Sleep/ Normal Meal
- Late Sleep/ Late Meal (Experimental): sleep 0330-1130 h, meals at 4.5, 8.5, 14.5, and 16 (snack) h after awakening
  Interventions: Behavioral: Late Sleep/ Late Meal

INTERVENTIONS:
Behavioral: Normal Sleep/ Normal Meal — The subject will be inpatient for 5 days, and sleep between the hours of 0000-0800 h, with meals at 1, 5, 11, and 12.5 (snack) h after awakening every day for 5 days. On night 3, we will insert a catheter in the participant's arm to facilitate multiple blood sampling overnight and the next day. On d 4, a frequently sampled i.v. glucose tolerance test (FSIVGTT) will be performed. A MTT will be performed at the scheduled lunch. At 1 h before dinner, participants will undergo fMRI scanning to assess neuronal responses to food stimuli and to examine functional connectivity with reward circuitry. On d 5, participants will be allowed to determine their own food intake at the scheduled meal and snack times. Participants will be discharged upon awakening on day 6.
  Arms: Normal Sleep/ Normal Meal
Behavioral: Normal Sleep/ Late Meal — The subject will be inpatient for 5 days and sleep between the hours of 0000-0800 h,with controlled meals at 4.5, 8.5, 14.5, and 16 (snack) h after awakening. On night 3, we will insert a catheter in the participant's arm to facilitate multiple blood sampling overnight and the next day. On d 4, at the scheduled breakfast time, a frequently sampled i.v. glucose tolerance test (FSIVGTT) will be performed. A MTT will be performed at the scheduled lunch. At 1 h before dinner, participants will undergo fMRI scanning to assess neuronal responses to food stimuli and to examine functional connectivity with reward circuitry. On d 5, participants will be allowed to determine their own food intake at the scheduled meal and snack times. Participants will be discharged upon awakening on day 6.
  Arms: Normal Sleep/ Late Meal
Behavioral: Late Sleep/ Normal Meal — The subject will be inpatient for 5 days, and sleep between the hours of 0330-1130 h, with controlled meals at 1, 5, 11, and 12.5 (snack) h after awakening. On night 3, we will insert a catheter in the participant's arm to facilitate multiple blood sampling overnight and the next day. On d 4, at the scheduled breakfast time, a frequently sampled i.v. glucose tolerance test (FSIVGTT) will be performed. A MTT will be performed at the scheduled lunch. At 1 h before dinner, participants will undergo fMRI scanning to assess neuronal responses to food stimuli and to examine functional connectivity with reward circuitry. On d 5, participants will be allowed to determine their own food intake at the scheduled meal and snack times. Participants will be discharged upon awakening on day 6.
  Arms: Late Sleep/ Normal Meal
Behavioral: Late Sleep/ Late Meal — The subject will be inpatient for 5 days, and sleep between the hours o 0330-1130 h, with controlled meals at 4.5, 8.5, 14.5, and 16 (snack) h after awakening. On night 3, we will insert a catheter in the participant's arm to facilitate multiple blood sampling overnight and the next day. On d 4, at the scheduled breakfast time, a frequently sampled i.v. glucose tolerance test (FSIVGTT) will be performed. A MTT will be performed at the scheduled lunch. At 1 h before dinner, participants will undergo fMRI scanning to assess neuronal responses to food stimuli and to examine functional connectivity with reward circuitry. On d 5, participants will be allowed to determine their own food intake at the scheduled meal and snack times. Participants will be discharged upon awakening on day 6.
  Arms: Late Sleep/ Late Meal

SUMMARY:
This study will test the hypothesis that a late sleep (Ls) and/or late meal (Lm) behavioral pattern, with equal sleep duration, will promote positive energy balance and insulin resistance (IR).

DETAILED DESCRIPTION:
Sleeping patterns affect aspects of metabolism that may impact obesity risk; our lab is interested in studying whether sleep patterns play a role in the development of obesity. Individuals with late bedtimes and late rise times tend to have greater food intake which includes more fast food and sugar-sweetened beverages, less fruits and vegetables [1], larger portions, and later eating times [2] than those with earlier bedtimes. This sleeping pattern is highly prevalent: ~15 million Americans work on shifts other than regular day hours [3] and others subject themselves to 'social jetlag' (time difference between the middle of the sleep episode [midpoint of sleep] on work days and non-work days, similar to travel across time zones) [4]. The shift in sleep and meal times associated with these lifestyles results in misalignment of sleep and eating behaviors with the circadian clocks. These clocks, located in the brain and organs throughout the body, regulate metabolism and behavior and are affected by sleep and feeding. Disruption of clock genes in individual organs may be in part responsible for metabolic dysregulation [5]. Altering the coordination of sleep and meal timing may affect food reward valuation (brain) and metabolism (peripheral organs) to promote obesity and IR, observed more frequently in shift workers. This is the focus of this randomized, crossover, controlled study of 4 phases:

* Normal sleep (Ns; 0000-0800 h), Normal meals (Nm=meals at 1, 5, 11, and 12.5 h after awakening)=Ns/Nm
* Normal sleep (Ns; 0000-0800 h), Late meals (Lm=meals at 4.5, 8.5, 14.5, and 16 h after awakening)=Ns/Lm
* Late sleep (Ls; 0330-1130 h), Normal meals (Nm=meals at 1, 5, 11, and 12.5 h after awakening)=Ls/Nm
* Late sleep (Ls; 0330-1130 h), Late meals (Lm=meals at 4.5, 8.5, 14.5, and 16 h after awakening)=Ls/Lm Aim 1: To determine whether Ls and/or Lm, in individuals with habitual normal sleep duration and timing, alters one or both sides of energy balance, i.e. food intake and energy expenditure (EE), relative to Ns and Nm.
* Hypothesis 1: (a) Ls and Lm will have independent and interactive effects on food intake and EE. Intake at an ad libitum test meal and during a 24 h period, measured after 3 d of each intervention, will be greater during Ls and Lm, and this will be enhanced when Ls and Lm are combined, compared to Ns and Nm. (b) Resting metabolic rate (RMR) will be lower during the Ls and Lm phases, and this will be further reduced when Ls and Lm are combined compared to the Ns and Nm phases (Ns/Nm<Ls/Nm≤Ns/Lm<Ls/Lm).

Aim 2: To determine whether neuronal responses to food stimuli in brain regions related to reward value explain differences in food intake.

• Hypothesis 2: (a) Increased brain activity in response to visual presentation of food stimuli, using functional magnetic resonance imaging (fMRI), will be seen in Ls and Lm compared to Ns and Nm in the insula and the orbitofrontal cortex. Enhanced neuronal activity in response to foods will be most pronounced in the Ls/Lm phase (Ns/Nm<Ls/Nm≤Ns/Lm<Ls/Lm). (b) Neuronal responses to food stimuli will be related to pre-test neuropeptide Y (NPY), hypocretin-1, and subsequent food intake.

Exploratory Aim 3: To determine whether meal or sleep timing affect glucose homeostasis and appetite-regulating hormones.

• Hypothesis 3: Ls and Lm will result in lower insulin sensitivity (frequently sampled i.v. glucose tolerance test [FSIVGTT] and meal tolerance test [MTT]) than Ns and Nm (Ns/Nm>Ls/Nm≥Ns/Lm>Ls/Lm). Sleep and meal timing will have independent and interactive effects on the 24-h pattern of hormones regulating food intake (lower leptin and glucagon-like peptide-1 [GLP-1]; higher ghrelin, NPY and hypocretin-1).

ELIGIBILITY:
Inclusion Criteria:

* Participants free of any current and past sleep and psychiatric disorders, including eating disorders (ex.anorexia, bulimia, night eating syndrome)
* Participants will not have diabetes and will normally consume a meal within 1 h after awakening at least 5 times/wk
* Participants with normal scores on the Pittsburgh Quality of Sleep Questionnaire [78] (global score <5) and Epworth Sleepiness Scale [79] (score <10), no indication of sleep apnea (Berlin Questionnaire) [80], sleep disorders (Sleep Disorders Inventory Questionnaire) [81], depression (Beck Depression Inventory II) [82], significant delayed or advanced sleep phase (Composite Scale of Morningness/Eveningness) [83], and involuntary sleep movement, by self-report.

Exclusion Criteria:

* Smokers (smoking any cigarettes or ex-smokers <3 y)
* Non-day and rotating shift workers
* Persons who plan to travel across time zones within 4 wk of the study
* Persons with a history of drug and alcohol abuse, drowsy driving, or excessive caffeine intake (>300 mg/d)
* Persons with recent weight change or who actively participated in a diet or weight loss program in the previous 3 mo.
* Individuals with a neurologic condition that may disrupt the procedures will be excluded
* Persons with low hematocrit (<30%) due to the high blood sampling protocol *Women who are pregnant or <1 y post-partum
* Individuals with contraindications for fMRI

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Food Intake | 24 h
  Energy, fat, protein, carbohydrate, sugar, fiber intakes by weighed intake measures

SECONDARY OUTCOMES:
Neuronal response | 1 h
  fMRI assessment of neuronal responses to food vs non-food stimuli and during the resting state
Cardio-metabolic risk profile | 1 day
  Frequently sampled i.v. glucose tolerance test; meal tolerance test (glucose and insulin) pattern of hormones regulating food intake (lower leptin and GLP-1; higher ghrelin, NPY and hypocretin-1

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- New York Nutrition Obesity Research Center, New York, New York, United States